CLINICAL TRIAL: NCT03436784
Title: The Effect of Supplemental Nutrition Assistance Program-Education on the Dietary Intake of Low-income Indiana Participants
Brief Title: The Indiana SNAP-Ed Long-term Study Sequel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Eicher-Miller, Assistant Prof. of Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1507016295
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Nutrient Intake Inadequacy

STUDY DESIGN:
Intervention Model Description: Parallel-arm intervention with inactive control group and intervention group
Who Masked: Participant
Masking Description: Participants who were recruited at the same time and location were assigned to the same treatment group to prevent knowledge of different treatment groups in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants who met eligibility requirements and agreed to be randomly allocated to a treatment group. The control group participants received no lessons. Control group participants received the same study assessments at the same timepoints as the intervention group. The control group participants may have had limited contact with the nutrition educators only to update contact information, to set or remind of appointments to complete study assessments, or to receive non-nutrition or non-resource management resources.
- Intervention Group (Experimental): Participants who met eligibility requirements and agreed to be randomly allocated to a treatment group.The Intervention group participants received lessons from the nutrition educators, completed the same study assessments at the same timepoints as the control group, and may have had additional interaction with the nutrition educators in accordance with normal Indiana SNAP-Ed protocol.
  Interventions: Behavioral: Indiana SNAP-Ed

INTERVENTIONS:
Behavioral: Indiana SNAP-Ed — First four Indiana SNAP-Ed nutrition education lessons served as the intervention
  Other Names: Small Steps to Health Curriculum
  Arms: Intervention Group

SUMMARY:
The goal of the study is to determine the immediate and long-term effects of SNAP-Ed on the dietary intake of participants.

DETAILED DESCRIPTION:
The goal of this study is to determine the efficacy of SNAP-Ed to improve the immediate and long-term dietary quality (using the Healthy Eating Index (HEI)), BMI (measured height and weight), and food security (using the 18-item US HFSSM) and how the provision of SNAP-Ed with the presence of other characteristics can mediate improvement in these outcomes. The hypothesis of this study is that dietary quality and food security will improve and BMI will remain steady over the short-term, and these improvements will be maintained over a 1-year, or "long-term", time frame in participants receiving SNAP-Ed compared to those not receiving SNAP-Ed. Results may be used as a basis for changes to the program or policies relevant to SNAP-Ed and other nutrition education programs throughout the US.

NEP educators are considered key personnel because they will have direct contact with study participants; however, they will not have any part in data entry, analysis, or dissemination of study results. NEP educators, employees of Purdue University Extension, across Indiana will help facilitate the study. NEP educators have completed CITI training as a requirement for employment through Purdue University Extension. Before recruiting study participants, participating NEP educators will attend training sessions facilitated by the co-investigators of the study. The training sessions will include instructions on how to interact with participants; answer questions related to the study; and protocol for administering surveys, measuring height and weight, keeping participant information private, and the use of identification numbers. The study goals and hypothesis will not be shared with the NEP educators in order to keep their work with the participants as unbiased as possible.

NEP educators will recruit study participants who are interested in participating in NEP. The details of recruitment are described in Section D. A screening survey determining eligibility will be administered in addition to an explanation of consent. After completion of the screening survey and consent process, NEP educators will randomize participants into one of two groups: control or experimental. The NEP educators will be assigned a random number using Excel and then listed in order from least to greatest according to their random number. The first half of the NEP educators will assign their first recruited participants to the experimental group. After the first assignment, they will alternate assigning participants to either study group in an "every other" participant fashion. The second half of the NEP educators will assign their first recruited participants to the control group. After the first assignment, they will also alternate assigning participants to either study group in an "every other" participant fashion. The control group will wait 1 year from taking the second survey before starting NEP lessons. The experimental group will start NEP lessons immediately. Participants in the experimental group must take at least the first 4 NEP lessons within a time period of 4 to 10 weeks. The NEP SNAP-Ed curriculum includes 10 lessons, and participants may take the additional 6 lessons if desired.

All participants will complete three 30 minute surveys throughout the study. Surveys will be administered by NEP educators using the Qualtrics Offline Application on their program-provided iPads or paper surveys. The first survey will be administered upon enrollment in the study. Participants in the experimental group will take the second survey after they have completed the first 4 lessons between 4 and 10 weeks after enrollment in the study. Control participants will take the second survey after 4 to 10 weeks with no lessons. Since participants will be recruited on a rolling basis, they will take surveys at different times within a designated time period. The third survey will be administered to both groups 1 year after the second survey. Surveys are comprised of the US Household Food Security Survey Module from the United States Department of Agriculture Economic Research Service, questions querying household and individual level characteristics, and the Indiana Food and Nutrition Program Evaluation Tool.

Participants will also complete two 24-hour dietary recalls using the Automated Self-Assisted 24-hour recall (ASA-24) and one food frequency questionnaire (FFQ) using the Diet History Questionnaire II (DHQ II) at each data collection time point. Both instruments are online and complementary dietary assessment tools created by the National Cancer Institute and have a respondent and researcher website. Results will be analyzed by the researchers using the researcher website. One dietary recall and the FFQ may be administered by the NEP Educators immediately following the in person survey, or a link to complete the dietary recall and FFQ online will be emailed to the participant within 2 days, or the participant can request to complete the dietary recalls and FFQ over the phone with the co-investigators at Purdue within 7 days after completing the survey. A script will be provided for the Purdue researchers to administer the dietary recalls and FFQ. The completion of the dietary recalls and the FFQ is necessary to perform complex modeling techniques for estimating usual dietary intake. The program that administers the dietary recalls assists participants through the recall process using an animated guide with audio and visual cues. Previous research has shown that the majority of Indiana SNAP-Ed participants have a computer with high-speed Internet connection in their home or residence. Participants without email, without access to a computer with internet, or with limited computer skills will be instructed to complete the assessments via telephone with assistance from researchers. If assistance from researchers is needed via telephone, participant identifying information will not be collected at that time. Participants will be identified only by their participant identification number, which they will receive upon enrollment in the study. Participants will provide days and time frames over the following week when they will be available to complete the dietary assessments over the phone with Purdue researchers. In addition, participants may call the co-investigator's Purdue office phone number any time after the survey for assistance with completing the dietary assessments. If the first dietary recall and FFQ have not been completed within 4 days after the survey, researchers will call the participant no more than once per day to complete the first dietary recall and FFQ over the phone at that time or to set up appointments to complete the dietary recalls and FFQ over the phone with researchers within the 7 days after completing the in person survey. The second dietary recall should be completed 24 hours after the first dietary recall at the earliest but before 9 days after completing the in person survey. Participants will have the same options as described above to complete the second dietary recall.

In addition to the survey, dietary recalls, and FFQ, NEP educators will take height and weight measurements on each participant at each assessment time point. Weights will be measured using the SECA 869 mobile medical flat scale with remote display. Heights will be measured using the SECA 213 mobile stadiometer. This weight scale and stadiometer are research grade measurement tools. Height and weight measurements will be taken following the Centers for Disease Control and Prevention (CDC) National Health and Nutrition Examination Survey (NHANES) anthropometry manual guidelines. Height and weight measurements will be completed in a private setting or privacy screens will be used. Only the NEP educators will be able to see the measurements. Three measurements will be taken at each assessment time point in order to calculate an average. Participants will be allowed to know their measurements upon request at the time of measurement. Researchers will use these measurements to calculate BMI.

An in person survey, two dietary recalls, one FFQ, and height and weight measurements will be completed for each participant at each of the three assessment time points. The first and third assessments will cover a reference period the past 12 months, while the second assessment will cover the past 30 days. Participants randomized to the control group will be provided the opportunity to complete the SNAP-Ed program at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* an interest in taking SNAP-Ed lessons
* willingness to wait 1 year to start FNP lessons
* eligibility for SNAP
* age of at least 18 years
* the household located in Indiana
* ability speak and read English
* willingness to complete three 45 minute surveys and up to 2 dietary recalls and a food frequency questionnaire at the designated time intervals
* willingness to stay in touch with research staff during the study period
* no previous participation in NEP lessons within the last year

Exclusion Criteria:

- pregnant women were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Long-term Change in Dietary Intake | Baseline assessments were completed upon recruitment and 1-year follow-up assessments were completed approximately 1 year after baseline assessments
  The Healthy Eating Index-2010 was used to characterize diet quality from National Cancer Institute Automated Self-Administered 24-hour Dietary Recall Tool

SECONDARY OUTCOMES:
Long-term Change in Nutrient Intake | Baseline assessments were completed upon recruitment and 1-year follow-up assessments were completed approximately 1 year after baseline assessments
  Mean Usual Intake was determined from National Cancer Institute Automated Self-Administered 24-hour Dietary Recall Tool
Long-term Change in Household Food Security | Baseline assessments were completed upon recruitment and 1-year follow-up assessments were completed approximately 1 year after baseline assessments
  Food security was measured by 18-item US Household Food Security Survey Module at baseline and 1-year follow-up assessment time points

OTHER OUTCOMES:
Body Mass Index (BMI) | Baseline assessments were completed upon recruitment and 1-year follow-up assessments were completed approximately 1 year after baseline assessments
  SNAP-Ed paraprofessionals measured height and weight to calculate BMI

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Eicher-Miller, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT03436784/Prot_003.pdf
  • Statistical Analysis Plan (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT03436784/SAP_005.pdf
  • Informed Consent Form (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT03436784/ICF_004.pdf